CLINICAL TRIAL: NCT02570620
Title: Apport de l'échographie du Col Dans l'évaluation du Délai Induction Accouchement (DIA) Chez Des Patientes à Score de Bishop défavorable après déclenchement Par Dinoprostone Intravaginal
Brief Title: Contribution of Ultrasonography in the Evaluation of Cervical Induction-delivery Time
Acronym: ECOLDIA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PHRI09-JP/ECOLDIA
Record Dates: First submitted 2015-10-02; First posted 2015-10-07 (Estimated); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Delivery Uterine; Birth; Induced

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Observational cohort of patients (Experimental): Patients will benefit from an ultrasonography of the cervix through endovaginal before induction of prostaglandins
  Interventions: Device: Ultrasonography of the cervix

INTERVENTIONS:
Device: Ultrasonography of the cervix

SUMMARY:
Study of the contribution of ultrasound measurements of the uterine cervix related to the calculation of Bishop score. Evaluation of the period between cervical induction and delivery. Study of ultrasound data to improve the care of these patients requiring induction.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Single pregnancy to term (> 37 weeks) in cephalic presentation
* Bishop score on the day of inclusion equal to 4.5 or 6
* Medical indication in accordance with professional recommendations of the April 2008 HAS.

Exclusion Criteria:

* Cicatricial uterus
* Placenta previa
* Parity > 3 (more than 3 previous deliveries > 22 weeks)
* History of cone biopsy and strapping
* Known fetal malformation
* Known allergy to prostaglandins
* Woman under guardianship

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 342 (Actual)
Dates: Start 2010-09; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Time in hours between induction of prostaglandins and delivery | On the day of inclusion after induction of prostaglandins. In relation to the time of delivery.
  Delivery whether a vaginal delivery or cesarean

CONTACTS AND LOCATIONS:
Overall Officials: Jérôme POTIN, Principal Investigator — University Hospital, Tours
Locations (3):
- France (3):
  - University Hospital of Nantes, Nantes
  - Hospital of Orleans, Orléans
  - University Hospital of Tours, Tours

REFERENCES:
- [Result] Arthuis C, Potin J, Winer N, Tavernier E, Paternotte J, Ramos A, Perrotin F, Diguisto C. Contribution of ultrasonography to the prediction of the induction-delivery interval: The ECOLDIA prospective multicenter cohort study. J Gynecol Obstet Hum Reprod. 2021 Dec;50(10):102196. doi: 10.1016/j.jogoh.2021.102196. Epub 2021 Jul 10. PMID 34256166